CLINICAL TRIAL: NCT06794775
Title: SWE-NEO: Swedish NeoAdjuvant Trial Comparing Anti-PD-1 Monotherapy to Combined Anti-CTLA-4/Anti-PD-1 Blockade in Resectable Stage III Melanoma
Brief Title: SWE-NEO: Swedish NeoAdjuvant Trial Comparing Monotherapy to Combined Immunotherapy in Resectable Stage III Melanoma
Acronym: SWE-NEO
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hildur Helgadottir (Other)
Responsible Party: Sponsor-Investigator, Hildur Helgadottir, Oncology consultant, Karolinska University Hospital
Organization: Karolinska University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SWE-NEO Trial
Record Dates: First submitted 2025-01-16; First posted 2025-01-27 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Malignant Melanoma Stage III
Keywords: Immune checkpoint inhibitors; Nivolumab; Ipilimumab; Neoadjuvant; anti-PD-1; anti-CTLA-4
MeSH Terms: conditions — Melanoma | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PD-1 inhibitor monotherapy (Active Comparator): Monotherapy with Nivolumab
  Interventions: Drug: Nivolumab
- PD-1/CTLA-4 inhibitor combination therapy (Experimental): Combination therapy with Nivolumab and Ipilimumab
  Interventions: Drug: Nivolumab + Ipilimumab

INTERVENTIONS:
Drug: Nivolumab — Adjuvant monotherapy with Nivolumab
  Arms: PD-1 inhibitor monotherapy
Drug: Nivolumab + Ipilimumab — Adjuvant combination therapy with Nivolumab and Ipilimumab
  Arms: PD-1/CTLA-4 inhibitor combination therapy

SUMMARY:
At present two studies (SWOG S1801 and NADINA) have demonstrated superiority when using neoadjuvant treatment compared to adjuvant treatment only, but no studies have compared PD-1 monotherapy (SWOG 1801 regimen) to the PD-1/CTLA-4 combination (NADINA regimen) therapy. The SWE-NEO study aims to compare these two regimens, where the PD-1/CTLA-4 combination is potentially more effective, but also associated with more side effects.

DETAILED DESCRIPTION:
A phase III randomized controlled multicenter open-label trial. Patients will be randomized after a diagnosis of resectable stage III melanoma to have either two courses of CTLA-4 and PD-1 inhibitor combination therapy or PD-1 inhibitor monotherapy, before the pre-planned operation. In both arms, adjuvant treatment with a PD-1 inhibitor or with BRAF+MEK inhibitors in patients with a BRAF V600E mutation, will be given only to patients with no major pathological response in the operated tumor, with PD-1 inhibitor, or with BRAF+MEK inhibitors in patients with BRAF V600E mutation. Active follow-up will be performed for 3 years from surgery and followed for survival up until 10 years. Sequential blood and tumor samples will be collected for biomarker analyses.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be at least 18 years of age.
2. Can provide a signed informed consent as described in the protocol, including compliance with the requirements and restrictions listed in the ICF and in this protocol.
3. World Health Organization (WHO) Performance Status 0 or 1.
4. Patients must have

   1. Histologically or cytologically confirmed Stage III melanoma. In the case of in-transit metastases (with or without lymph node metastases)' ≤3 resectable in-transit metastases are allowed.
   2. Patients with cutaneous, acral, or unknown primary melanomas are eligible for enrollment.
   3. Resectable tumors are defined as having no significant vascular, neural or bony involvement. Only patients where a complete surgical resection with tumor-free margins can safely be achieved are defined as resectable.
5. Female patient of childbearing potential should have a negative urine or serum pregnancy test within 72 hours prior to receiving the first treatment. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
6. Female patients of childbearing potential must be willing to use a highly effective method of contraception, for the course of the study through 150 days after the last dose of study medication. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject. Highly effective methods of contraception include one or more of the following:

   1. male partner who is sterile (vasectomised) prior to the female study subject's entry into the study and is the sole sexual partner for the female subject;
   2. hormonal (oral, intravaginal, transdermal, implantable or injectable)
   3. an intrauterine hormone-releasing system (IUS)
   4. an intrauterine device (IUD) with a documented failure rate of < 1%.
7. Male patients of childbearing potential must agree to use an adequate method of contraception, starting with the first dose of study therapy through 150 days after the last dose of study therapy. Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject. A unique female sexual partner must postmenopausal, permanently sterilized (e.g. hysterectomy or tubal ligation), or use a highly effective method of contraception.
8. No other malignancies, except if treated with curative intent and with a cancer-related life expectancy of more than 5 years.
9. No prior immunotherapy targeting CTLA-4, PD-1 or PD-L1.
10. No prior targeted therapy targeting BRAF and/or MEK.

Exclusion Criteria:

1. Unresectable melanoma
2. Uveal/ocular or mucosal melanoma
3. Any serious or uncontrolled medical conditions that, in the investigator's opinion, may increase the risk associated with study participation or study drug administration, impair the ability of the subject to receive protocol therapy, or interfere with the interpretation of study results .
4. Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
5. Women who are pregnant or breastfeeding.
6. Any condition that potentially hamper compliance with the study protocol and follow-up schedule; those conditions should be discussed with the subject before registration in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2025-07-10 (Actual); Primary Completion 2032-04-15 (Estimated); Study Completion 2032-04-15 (Estimated)

PRIMARY OUTCOMES:
Event-free survival (EFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  Event-free survival (EFS), defined as time from randomization to melanoma progression (irresectable stage III or stage IV disease), melanoma recurrence, or death from any cause (treatment-related, melanoma related or any other).

SECONDARY OUTCOMES:
Relapse-free survival (RFS) | From date of surgery until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  Relapse-free survival (RFS), defined as time between date of surgery and date of melanoma recurrence, treatment-related death or melanoma-related death, whichever occurs first.
Distant metastasis-free survival (DMFS) | From date of randomization until the date of first documented distant metastasis or date of death from any cause, whichever came first, assessed up to 60 months
  Distant metastasis-free survival (DMFS), defined as time between date of randomization and date of first distant metastasis, treatment-related death or melanoma-related death, whichever occurs first.
Overall survival (OS) | From date of randomization until the date of death from any cause, assessed up to 60 months
  Overall survival (OS), defined as time between date of randomization and date of death.
Major pathological response (MPR) | Start of neoadjuvant therapy to end of neoadjuvant therapy, up to approximately two months
  Major pathological response (MPR) (≤10% viable tumor cells), difference in MPR between combined ICI and monotherapy, central review of all surgical specimens by three expert melanoma pathologists.
Correlation of pathologic response to RFS, DMFS, and OS | From end of neoadjuvant therapy until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  Correlation of pathologic response in each arm to RFS, DMFS, and OS.
Correlation of response to RFS, DMFS, and OS | From end of neoadjuvant therapy until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  Correlation of radiological and clinical response evaluation to RFS, DMFS, and OS.
Proportion of patients having surgery according to plan | From start of neoadjuvant therapy to date of surgery, assessed up to 6 months
  Number of patients having surgery according to plan (within 10 weeks from first neoadjuvant course).
Surgical complication rates | From surgery to date of any postoperative complication, assessed up to 3 months post surgery
  Surgical complication rates according to Clavien-Dindo surgical classification.
Frequency of treatment-related adverse events (AEs) | From start of neoadjuvant therapy up to 1 year after last treatment
  Frequency of all grade and grade 3-5 treatment-related adverse events (AEs) according to CTCAE 5.0.

OTHER OUTCOMES:
Correlation of different biological markers with treatment efficacy and safety | From start of neoadjuvant therapy to last blood/tumour sample taken, until the date of first documented progression, assessed up to 60 months
  The explorative endpoints of this trial are:
  Correlation of different biological markers analyzed from sequential blood and tumor samples with treatment efficacy and safety.

CONTACTS AND LOCATIONS:
Locations (3):
- Sweden (3):
  - Sahlgrenska University Hospital, Gothenburg
  - Skane University Hospital, Lund
  - Karolinska University Hospital, Stockholm